CLINICAL TRIAL: NCT05743036
Title: A Phase 1/2, Open-Label, Multi-Center Study of ZN-c3 Administered in Combination With Encorafenib and Cetuximab in Adults With Metastatic Colorectal Cancer
Brief Title: ZN-c3 in Adult Participants With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to change in therapeutic landscape.
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-016; Z0011001 (Other: Pfizer)
Record Dates: First submitted 2023-01-26; First posted 2023-02-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; CRC; BRAF V600E
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Participants will receive different doses of ZN-c3 in combination with different doses of Encorafenib and a fixed dose of Cetuximab
  Interventions: Drug: ZN-c3; Drug: Encorafenib; Drug: Cetuximab
- Dose Expansion (Experimental): Participants will receive recommended dose of ZN-c3 and encorafenib as determined in dose escalation phase in combination with cetuximab
  Interventions: Drug: ZN-c3; Drug: Encorafenib; Drug: Cetuximab

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 tablet by mouth, in combination with encorafenib
Drug: Encorafenib — Encorafenib capsule by mouth, in combination with ZN-c3
  Other Names: BRAFTOVI®
Drug: Cetuximab — Infusion
  Other Names: ERBITUX®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and potential clinical benefits of ZN-c3 administered in combination with encorafenib and cetuximab in adult participants with metastatic BRAF V600E mutant colorectal cancer previously treated with one or two treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic Stage IV colorectal adenocarcinoma.
* Documented evidence of a BRAF V600E mutation in tumor tissue or blood
* Presence of measurable disease per RECIST version 1.1 guidelines.
* Disease progression after 1 or 2 previous systemic regimens for metastatic disease
* Adequate bone marrow function
* Adequate hepatic and renal function

Exclusion Criteria:

* Documented clinical disease progression or radiographic disease progression during the screening period
* Leptomeningeal disease.
* Symptomatic brain metastasis.
* Presence of acute or chronic pancreatitis.
* Unable to swallow, retain, and absorb oral medications.
* Clinically significant cardiovascular diseases
* Evidence of active noninfectious pneumonitis.
* Evidence of active and uncontrolled bacterial or viral infection, within 2 weeks prior to start of any of the study interventions
* Participants with known positivity for HIV
* Active hepatitis B or hepatitis C infection
* Concurrent or previous other malignancy within 2 years of study entry
* Has had an allogeneic tissue/solid organ transplant
* Pregnant or females of childbearing potential who have a positive β-hCG laboratory test result within 14 days prior to enrollment or is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Phase - Incidence of Dose Limiting Toxicities (DLTs) | From Lead-in Day -1 to Cycle 1 Day 28
  DLTs defined as treatment-related AEs occurring within the first 29 days after the start of any study treatment that in the opinion of the investigator cannot be reasonably attributed to the participant's underlying disease, concomitant medications, or pre-existing conditions.
Dose Expansion Phase - Objective response rate (ORR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  ORR defined as the proportion of participants who achieves a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Investigator per RECIST Version 1.1.

SECONDARY OUTCOMES:
Dose Escalation Phase - Incidence and severity of adverse events (AEs) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 | From first dose of any study intervention through 28 days after the last dose of any study intervention
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Proportion of participants with dose interruptions due to AEs in Dose Escalation Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Proportion of participants with dose modifications due to AEs in Dose Escalation Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Proportion of participants with discontinuations due to AEs in Dose Escalation Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Dose Escalation Phase - Objective response rate (ORR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  ORR defined as the proportion of participants who achieved a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) per RECIST Version 1.1.
Dose Escalation Phase - Duration of Response (DOR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  DOR defined as the time from the date of first radiographic evidence of response (CR or PR) to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Dose Escalation Phase - Progression Free Survival (PFS) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  PFS defined as the time from the first dose to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Dose Escalation Phase - Disease Control Rate (DCR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  DCR defined as the proportion of participants with BOR of CR, PR, or stable disease (SD), per RECIST version 1.1.
Dose Escalation Phase - Time to Response (TTR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  TTR defined as the time from first dose to first radiographic evidence of response (CR or PR) per RECIST version 1.1.
Dose Escalation - ZN-c3 plasma exposure: AUC | From lead in day -1 visit through Cycle 1 Day 15
Dose Escalation - ZN-c3 plasma exposure: Cmax | From lead in day -1 visit through Cycle 1 Day 15
Dose Escalation - ZN-c3 plasma exposure: Tmax | From lead in day -1 visit through Cycle 1 Day 15
Dose Escalation - Encorafenib plasma exposure: AUC | From lead in day -1 visit through Cycle 1 Day 15
Dose Escalation - Encorafenib plasma exposure: Cmax | From lead in day -1 visit through Cycle 1 Day 15
Dose Escalation - Encorafenib plasma exposure: Tmax | From lead in day -1 visit through Cycle 1 Day 15
Dose Expansion Phase - Duration of Response (DOR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  DOR defined as the time from the date of first radiographic evidence of response (CR or PR) to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Dose Expansion Phase - Progression Free Survival (PFS) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  PFS defined as the time from the first dose to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Dose Expansion Phase - Disease Control Rate (DCR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  DCR defined as the proportion of participants with BOR of CR, PR, or stable disease (SD), per RECIST version 1.1.
Dose Expansion Phase - Time to Response (TTR) | From first dose of any study intervention every 8 weeks during treatment, up to 12 months
  TTR defined as the time from first dose to first radiographic evidence of response (CR or PR) per RECIST version 1.1.
Dose Expansion Phase - Incidence and severity of adverse events (AEs) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 | From first dose of any study intervention through 28 days after the last dose of any study intervention
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Proportion of participants with dose interruptions due to AEs in Dose Expansion Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Proportion of participants with dose modifications due to AEs in Dose Expansion Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Proportion of participants with discontinuations due to AEs in Dose Expansion Phase | From first dose of any study intervention through 28 days after the last dose of any study intervention
Dose Expansion - ZN-c3 in combination with combination with E+C plasma exposure: AUC | Lead in day 7
Dose Expansion - ZN-c3 in combination with combination with E+C plasma exposure: Cmax | Lead in day 7
Dose Expansion - ZN-c3 in combination with combination with E+C plasma exposure: Tmax | Day 7
Dose Expansion - Encorafenib in combination with ZN-c3 and cetuximab plasma exposure: AUC | Cycle 1 Day 15
Dose Expansion - Encorafenib in combination with ZN-c3 and cetuximab plasma exposure: Cmax | Cycle 1 Day 15
Dose Expansion - Encorafenib in combination with ZN-c3 and cetuximab plasma exposure: Tmax | Cycle 1 Day 15
Dose Expansion - ZN-c3 plasma exposure: AUC | Cycle 1 Day 15
Dose Expansion - ZN-c3 plasma exposure: Cmax | Cycle 1 Day 15
Tumor tissue BRAF V600E mutational status | From lead in day 1 visit through the last dose of any study intervention, up to 12 months

CONTACTS AND LOCATIONS:
Locations (27):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Alliance for Multispecialty Research, LLC, Merriam, Kansas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Germany (5):
  - Hämatologie- Onkologie im Zentrum MVZ GmbH, Augsburg, Bavaria
  - Klinikum der Universität München Großhadern, Munich, Bavaria
  - Muenchen Klinik Neuperlach, Klinik fuer Haematologie und Onkologie, Munich, Bavaria
  - Institut für Klinisch Onkologische Forschung, Frankfurt am Main, Hesse
  - DRK Kliniken Berlin - Köpenick, Berlin, State of Berlin
- Hungary (2):
  - Semmelweis University-Department of Internal Medicine and Oncology, Budapest, Budapest
  - Clinexpert Kft. Bugat Pal Korhaz, Gyöngyös
- Italy (5):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Europeo di Oncologia, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - AOUI Verona, Verona, Veneto
- Poland (4):
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Koszarowskiego, Opole, Opole Voivodeship
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat

IPD SHARING:
Plan to Share IPD: No